CLINICAL TRIAL: NCT03940092
Title: Sodium (23Na) MRI for Tumour Characterisation and Assessment of Therapy Response in Breast Cancer
Acronym: NaRNIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Fiona J Gilbert, Head of Department of Radiology; Consultant Radiologist, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 260281
Record Dates: First submitted 2019-04-30; First posted 2019-05-07 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathological analysis will be performed on diagnostic biopsies and tumour specimens from participating breast cancer patients. Immunohistochemical staining will be performed on histological samples to assess tumour vascularity, metabolism, and other markers of interest for correlation with imaging findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers: Healthy volunteers will be scheduled for an 23Na-MR examination
  Interventions: Other: MRI
- Breast cancer patients (primary surgery): Patients scheduled for primary surgery will undergo a single MR examination, involving 23Na-imaging prior to their planned surgery.
  Interventions: Other: MRI
- Breast cancer patients (neoadjuvant chemotherapy): Patients undergoing neo-adjuvant therapy will undertake up to two (2) combined PET/MR examinations with FDG. Examinations will be conducted at baseline and after 3-4 cycles of chemotherapy.
  Interventions: Other: PET/MRI

INTERVENTIONS:
Other: MRI — This is a prospective, non-randomised, exploratory study on healthy female volunteers (>18 years), and female patients (>18 years) diagnosed with primary breast cancer.
  Healthy volunteers will be scheduled for an 23Na-MRI examination.
  Patients scheduled for primary surgery will undergo an MR examination, involving 23Na-imaging prior to their planned surgery.
  Other Names: 23Na-MRI
  Groups: Breast cancer patients (primary surgery); Healthy Volunteers
Other: PET/MRI — Patients undergoing neo-adjuvant chemotherapy will undertake up to two (2) combined PET/MR examinations with FDG and 23Na-MRI
  Other Names: FDG-PET/MRI
  Groups: Breast cancer patients (neoadjuvant chemotherapy)

SUMMARY:
The scope of this study is the methodological development and optimisation of sodium MRI (23Na-MRI) protocols for breast cancer imaging. The study further proposes to utilise biomarkers obtained from 23Na-imaging (cell integrity), FDG-PET (metabolism), multi-parametric MRI (perfusion, vascularity, cellularity, morphology) to generate parameter maps specific for physiological processes in breast cancer.

DETAILED DESCRIPTION:
This is a prospective, non-randomised, exploratory study on ≤20 healthy female volunteers (>18 years), and ≤45 female patients (>18 years) diagnosed with primary breast cancer. Healthy volunteers (n≤20) will be scheduled to undergo an 23Na-MR examination. Patients scheduled for primary surgery (n≤30) will undergo a single MR examination, involving 23Na-imaging prior to their planned surgery. Immunohistochemical analysis will be performed on surgical tissue specimens to determine tissue markers of interest for correlation with the imaging findings. Patients undergoing neo-adjuvant therapy (n≤15) will undertake up to two (2) combined PET/MR examinations with FDG (18F-2-fluoro-2-deoxy-D-glucose) and 23Na-MRI. Patient imaging will occur at two time points prior to their planned surgery: (i) baseline (prior to initiation of treatment) and (ii) mid-treatment (after 3-4 cycles of chemotherapy). Histopathological analysis will be performed on pre-treatment biopsies for histological markers of interest for correlation with the imaging findings.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* Female, aged 18 years or above
* Participant is willing and able to give informed consent for participation in the study.

Patients

* Female, aged 18 years or above
* Pathologically confirmed primary breast cancer
* Tumour >1 cm diameter on mammography and/or ultrasound.

Exclusion Criteria for healthy volunteers and patients:

* Pregnant or lactating;
* History of serious breast trauma within past 3 months
* Implants known to be contraindicated at 3T MRI
* Significant or uncontrolled medical problems which according to the opinion of the Principal Investigator render the participant unsuitable for participation in the study
* Underlying conditions, including but not limited to medical or psychiatric conditions, which in the opinion of the Principal Investigator would preclude the participant from adhering to the study protocol or completing the study per protocol
* Lacking the capacity to provide informed consent.

Additional exclusion criteria for patients

* Has undergone chemotherapy or hormonal therapy for breast cancer in the previous 12 months
* Previous surgery or radiotherapy for breast cancer to the ipsilateral breast within the past 4 months
* Previous surgery for benign breast disease within the past 4 months
* History of kidney disease or known allergic reaction to gadolinium contrast agent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy female volunteers (n≤20), aged 18 years or above.
  Female patients (n≤45) aged 18 years or above, with pathologically confirmed primary breast cancer undergoing primary surgery or neo-adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Image quality of 23Na-MRI in the breast evaluated radiologically after each 23Na-MRI scan in healthy volunteers and patients. | Up to 2 years
  Development and optimisation of protocols for the imaging of intra and extracellular 23Na in breast cancer. Protocols will be developed on healthy volunteers and applied on cohorts of breast cancer patients

SECONDARY OUTCOMES:
Correlation of baseline 23Na-MRI with tissue markers of metabolism | Up to 2 years
  Correlation of baseline tissue sodium concentration as measured by 23Na-MRI with tissue markers of metabolism obtained from histopathological analysis of diagnostic biopsies/specimens
Change in 23Na-MRI measurements in breast cancer patients undergoing neo-adjuvant therapy | Up to 2 years
  Feasibility of measuring changes 23Na-MRI measurements in breast cancer patients undergoing neo-adjuvant therapy

OTHER OUTCOMES:
Correlate changes between 23Na-MRI measurements and changes in FDG-PET and multi-parametric proton-MR imaging | Up to 2 years
  Correlation of changes between 23Na-MRI measurements and changes in FDG-PET/multi-parametric proton-MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Gilbert, FRCR, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No